CLINICAL TRIAL: NCT01036087
Title: Phase II Study of Panitumumab, Nab-paclitaxel, and Carboplatin for Patients With Primary Inflammatory Breast Cancer (IBC) Without HER2 Overexpression
Brief Title: Panitumumab, Nab-paclitaxel and Carboplatin for HER2 Negative Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0372; NCI-2012-00935 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Inflammatory Breast Cancer; IBC; Primary breast carcinoma; HER2 negative overexpression; Panitumumab; Vectibix; Nab-paclitaxel; Paclitaxel; Abraxane; Carboplatin; Paraplatin; PNC; 5-fluorouracil; 5-FU; Adrucil; Efudex; Epirubicin; Ellence; Cyclophosphamide; Cytoxan; Neosar; FEC
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Panitumumab; 130-nm albumin-bound paclitaxel; Taxes; Albumin-Bound Paclitaxel; Carboplatin; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PNC + FEC (Experimental): PNC = Panitumumab + Nab-paclitaxel + Carboplatin, and
  FEC = 5-fluorouracil, epirubicin, and cyclophosphamide
  Interventions: Drug: Panitumumab; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Panitumumab — 2.5 mg/kg IV on Day 1 of Week 1 over 60 minutes, followed by 2.5 mg/kg weekly Weeks 2-12.
  Other Names: Vectibix
Drug: Nab-paclitaxel — 100 mg/m2 IV over 30 min on Day 1 of Weeks 2-13 over 30 minutes.
  Other Names: Paclitaxel (protein-bound); Abraxane; ABI-007
Drug: Carboplatin — AUC 2 IV over 30 min on Day 1 of Weeks 2-13 after completion of Abraxane through separate IV line.
  Other Names: Paraplatin
Drug: 5-Fluorouracil — 500 mg/m2 IV every 3 weeks, starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
  Other Names: 5-FU; Adrucil; Efudex
Drug: Epirubicin — 100 mg/m2 IV over 30 min every 3 weeks starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
  Other Names: Ellence
Drug: Cyclophosphamide — 500 mg/m2 IV every 3 weeks starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
  Other Names: Cytoxan; Neosar

SUMMARY:
The goal of this clinical research study is to learn how effective the combination of chemotherapy including both panitumumab, Abraxane (nab-paclitaxel), and carboplatin (PNC) and fluorouracil, epirubicin, and cyclophosphamide (FEC) used before surgery for the treatment of IBC is. The safety of PNC combination will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Panitumumab is designed to prevent or slow down the growth of tumor cells by blocking the proteins on the surface the cancer cell, called the epidermal growth factor receptor (EGFR).

Nab-paclitaxel is designed to kill tumor cells by binding a chemotherapy drug paclitaxel to albumin, a protein made by the liver. The albumin gets into the cancer cell and releases the paclitaxel directly to the tumor.

Carboplatin is designed to stop or slow cancer cells from growing by damaging the RNA or DNA (the genetic material of cells) that tells the tumor cells to grow.

5-fluorouracil, epirubicin, and cyclophosphamide each work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

Study Drug Administration:

On Day 1 of Week 1, you will receive panitumumab through a needle in your vein over 60 minutes.

After Week 1, you will receive a total of 4 cycles of PNC. Each cycle is 4 weeks.

During Cycles 1-3 (Weeks 2-13), you will receive PNC by vein once a week for 3 weeks, followed by a week of rest. You will receive PNC through a needle in your vein. The infusion will take 90 minutes.

During Cycle 4 (Week 14 to 17), you will receive PNC on Day 1 of Weeks 14 and 15. On Day 1 of Week 16, you will receive only carboplatin and nab-paclitaxel.

Starting on Day 1 of Week 18, you will receive FEC through a needle in your vein. The infusion will take 90 minutes. You will receive a total of 4 cycles, each 3 weeks long, over 12 weeks.

Surgery:

After you have completed both PNC and FEC treatments, you will have the standard of care surgery performed. You will be given a separate consent form to read and sign.

During surgery, breast tissue samples will be collected to identify tumors as routine procedure.

Study Visits:

Each week that you receive PNC or FEC therapy, before each dose of chemotherapy, blood (about 1 1/2 tablespoons) will be drawn for routine tests.

Before Week 2, an optional breast core biopsy will be performed to collect tumor samples for biomarker testing

On Week 2, every 4 weeks after that until the end of PNC, and again before FEC, the following tests and procedures will be performed before each dose of chemotherapy.

* You will have a physical exam, including measurement of your vital signs and weight, and breast exam.
* Blood (about 1 1/2 tablespoons) will be drawn for routine tests.
* You will be asked how well you are able to perform the normal activities of daily living (performance status).

During Weeks 2 and 9, and before FEC therapy, the study doctor will take pictures of both of your breasts.

Before FEC (after Cycle 4 of PNC) and again before surgery, the following tests and procedures will be performed:

* To check the status of the disease, imaging studies including mammogram, breast MRI, breast ultrasound, and digital photograph will be performed.
* You will have a physical exam, including vital signs, weight, and breast exam
* Blood (about 3 tablespoons) will be drawn for routine tests.
* You will be asked about any symptoms that you may have.
* The ECGs and ECHO/MUGA scans will be repeated, when the doctor thinks it is necessary.

This schedule may be changed if the study doctor thinks that it is necessary.

Length of the study:

You may remain on study treatment for up to 10 months. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

This is an investigational study. Panitumumab is FDA approved and commercially available for the treatment of EGFR-expressing metastatic colorectal cancer with disease progression. It's use in this study is considered to be investigational.

Nab-paclitaxel is FDA approved and commercially available for the treatment of breast cancer after the failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy. The use of Nab-paclitaxel in this study is considered to be investigational.

Carboplatin is FDA approved and commercially available for the treatment of IBC.

FEC is FDA approved for breast cancer in general, but not specifically for inflammatory breast cancer.

The use of PNC and FEC together before surgery is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of breast carcinoma. Pathologic evidence of dermal lymphatic invasion should be noted but not required.
2. Clinical diagnosis of IBC (presence of inflammatory changes in the involved breast, including diffuse erythema, heat, ridging, and peau d'orange).
3. >/= Age 18
4. ECOG performance status </= 1
5. Adequate hematologic function: Absolute neutrophil count (ANC) >/= 1.5 x 109/L, Platelet count >/= 100 x 109/L, Hemoglobin >/= 9.0 g/dL
6. Adequate cardiac function (LVEF >/= 45%)
7. Adequate Renal function: Creatinine (Cr) </= 1.5 mg/dL x ULN, Creatinine clearance (CrCl) >/= 50 mL/min calculated by the Cockcroft-Gault method as follows: Male creatinine clearance = (140 - age) x (weight in Kg) / (serum Cr x 72) Female CrCl = (140 - age) x (weight in Kg) x 0.85 / (serum Cr x 72)
8. Adequate Hepatic function: Aspartate aminotransferase (AST) </= 2.5 x ULN • Alanine aminotransferase (ALT) </= 2.5 x ULN • Alkaline phosphatase (Alp) </= 2.5 x ULN.Total bilirubin </=1.5 x ULN
9. Ability and willingness to sign an informed consent form for this protocol
10. If female of childbearing potential (women who are post-menopausal < 1 year, not surgically sterilized, or not abstinent), pregnancy urine test is negative, and agrees to be consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile prior to the female subject entry into the study and is the sole sexual partner for that female subject; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraception, or barrier methods, including diaphragm or condom with a spermicide.
11. Patients who have metastatic disease, if the metastatic sites are amendable for local therapy (i.e. radiation and/or surgery), and are candidates for breast surgery will be eligible,

Exclusion Criteria:

1. History of radiation or chemotherapy
2. HER2-positive breast carcinoma (IHC staining more than 3+ or HER2 gene amplification by FISH)
3. Recurrent breast cancer
4. History of other malignancies (except for cured non-melanomatous skin cancer or cured cervical carcinoma in situ, or malignancies with no evidence of disease and no treatment for >5 years)
5. Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
6. History of extensive interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of extensive interstitial lung disease on baseline chest CT scan
7. Patient with other significant medical or psychiatric condition that would make assessment of toxicity or efficacy difficult.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Peripheral neuropathy >= Gr II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Matsuda N, Wang X, Lim B, Krishnamurthy S, Alvarez RH, Willey JS, Parker CA, Song J, Shen Y, Hu J, Wu W, Li N, Babiera GV, Murray JL, Arun BK, Brewster AM, Reuben JM, Stauder MC, Barnett CM, Woodward WA, Le-Petross HTC, Lucci A, DeSnyder SM, Tripathy D, Valero V, Ueno NT. Safety and Efficacy of Panitumumab Plus Neoadjuvant Chemotherapy in Patients With Primary HER2-Negative Inflammatory Breast Cancer. JAMA Oncol. 2018 Sep 1;4(9):1207-1213. doi: 10.1001/jamaoncol.2018.1436. PMID 29879283
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2010- July 2015. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 47 participants were accrued and assessed for eligibility. 7 participants were ineligible and excluded ( 3 had HER2-positive disease, 2 had metastatic disease, and 2 did not receive financial approval for treatment.
Groups:
- PNC + FEC: PNC = Panitumumab + Nab-paclitaxel + Carboplatin, and
  FEC = 5-fluorouracil, epirubicin, and cyclophosphamide
  Panitumumab: 2.5 mg/kg IV on Day 1 of Week 1 over 60 minutes, followed by 2.5 mg/kg weekly Weeks 2-12.
  Nab-paclitaxel: 100 mg/m2 IV over 30 min on Day 1 of Weeks 2-13 over 30 minutes.
  Carboplatin: AUC 2 IV over 30 min on Day 1 of Weeks 2-13 after completion of Abraxane through separate IV line.
  5-Fluorouracil: 500 mg/m2 IV every 3 weeks, starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
  Epirubicin: 100 mg/m2 IV over 30 min every 3 weeks starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
  Cyclophosphamide: 500 mg/m2 IV every 3 weeks starting on Day 1 of Week 14 (4 cycles, each 3 weeks long, over 12 weeks).
Period: Overall Study
Arm/Group | PNC + FEC
Started | 40
Completed | 37
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | PNC + FEC
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 57 [23 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 11
  Postmenopausal | 29
Clinical N Category [Count of Participants; unit: Participants] — N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N1 | 20
    N2 | 4
    N3 | 16
Clinical TNM Stage at Presentation [Count of Participants; unit: Participants] — Clinical Stage for inflammatory breast cancer was determined by the presence of distant metastases at initial diagnosis. Stage III was confined to the regional area and stage IV had distant metastases. Stage IV was considered worse outcomes.
  Participants
    III | 36
    IV | 4
Nuclear Grade [Count of Participants; unit: Participants] — A low grade number (grade 1) usually means the cancer is slower-growing and less likely to spread. A high grade number (grade 3) means a faster-growing cancer that's more likely to spread. An intermediate grade number (grade 2) means the cancer is growing faster than a grade 1 cancer but slower than a grade 3 cancer.
  Participants
    Grade 2 | 13
    Grade 3 | 27
Primary Tumor Subtype [Count of Participants; unit: Participants]
  HR Positive HER2 negative | 21
  HR Negative HER2 negative | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved Pathologic Complete Response (CR)
Description: Pathologic complete response was defined as absence of invasive carcinoma in the breast, axillary lymph nodes, and skinand absence of tumor emboli within the surgical field.
Time Frame: Assessed after 14 weeks (following PNC and FEC preoperative chemotherapy treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | PNC + FEC
Number analyzed (Participants) | 40
Participants | 11

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: AEs were graded according to the National Cancer Institute's Common Terminology Criteria (CTCAE), version 3.0. All AEs (>/=2 non-hematological and >/=3 hematological AEs) occurring after informed consent signing observed by the investigator or reported by the subject whether or not attributed to investigational product. Full AE reporting can be found in the Adverse Event Section.
Time Frame: Before each cycle of Panitumumab, nab-paclitaxel and carboplatin (PNC) & fluorouracil, epirubicin and cyclophosphamide (FEC) until 30 days after the last dose of drug, an average of 8 months, unless the participant withdraw consent.
Measure: Count of Participants; unit: Participants
Arm/Group | PNC + FEC
Number analyzed (Participants) | 40
Participants
  >/=2 non-hematological AEs | 36
  >/=3 hematological AEs | 26

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdrew consent, an average of 8 months.
Arm/Group | PNC + FEC
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 15/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNC + FEC (N=40)
Bleeding per rectum (Gastrointestinal disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Delirium (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
MDS (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Sycope (Nervous system disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vulvar abscess (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PNC + FEC (N=40)
Leukopenia (Blood and lymphatic system disorders) | 9
Neutrophil count decreased (Blood and lymphatic system disorders) | 26
Hemoglobin decreased (Blood and lymphatic system disorders) | 7
Platelet count decreased (Blood and lymphatic system disorders) | 8
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 33
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 23
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 23
Hypersensitivity (General disorders) | 2
Hand-and-foot syndrome (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 7
Infection (Infections and infestations) | 7
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Urinary tract infection (Renal and urinary disorders) | 4
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT01036087/Prot_SAP_000.pdf